CLINICAL TRIAL: NCT07076628
Title: Incidence of Respiratory Depression of Remimazolam Compared With Propofol for Monitored Anesthesia Care During Hysteroscopy
Brief Title: Respiratory Depression of Remimazolam vs. Propofol for Monitored Anesthesia Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Junyong In, MD, PhD, Professor, DongGuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: J In 2021-1
Record Dates: First submitted 2022-02-02; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Propofol; Remimazolam; Hysteroscopic Surgery; Respiratory Insufficiency; Hemodynamics Instability
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Propofol; remimazolam

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled to one of the two drug groups with randomization.
Who Masked: Participant, Investigator
Masking Description: Care giver will notice which drug will be given to the patients because of the color (White vs clear) and infusion doses of the drugs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol group (Active Comparator): Propofol infusion with remifentanil for hysteroscopic surgery
  Interventions: Drug: Propofol
- Remimazolam group (Active Comparator): Remimazolam infusion with remifentanil for hysteroscopic surgery
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Propofol — Propofol infusion with remifentanil
  Arms: Propofol group
Drug: Remimazolam — Remimazolam infusion with remifentanil
  Arms: Remimazolam group

SUMMARY:
The comparison of incidence of respiratory depression between remimazolam and propofol under monitored anesthesia care for hysteroscopic surgery

DETAILED DESCRIPTION:
* Non-invasive blood pressure, electrocardiogram, and oxygen saturation sensors are attached.

  * Wear an oxygen mask (5L per minute), and place the sampling line for end-tidal carbon dioxide partial pressure measurement inside the nose.

    * Check the randomization table to determine the drug to be administered, and prepare propofol or remimazolam accordingly.

      * Record the baseline values (0 min).

        * Start administration of Remifentanil.

          ⑥ Administer anesthesia to adjust the maintenance dose to reach a sedation level of 2 or less on the MOAA/S scale.

          ⑦ Adjust the remifentanil dose according to the patient's response

          ⑧ When the target sedation level is reached, the surgical preparation process and surgery begin, and the study variables are observed and recorded at 5-minute intervals.

          ⑨ Stop drug administration upon end of surgery.

          ⑩ After confirming proper recovery of consciousness and spontaneous breathing, leave the recovery room.

          ⑪ Before leaving the recovery room, check the complete recovery and investigate the patient's satisfaction with anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS 1-2
* Elective hysteroscopic surgery under monitored anesthesia care
* No drug abuse history

Exclusion Criteria:

* BMI > 30 kg/m2
* Hepatic or renal insufficiency
* Alcohol abuse
* Respiratory, hemodynamic compromise, or diseases
* History of general/regional anesthesia during the last month
* A patient who is taking sedatives or analgesics
* Under the investigator's judgment

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — with gynecologic surgery
Enrollment: 76 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Respiratory insufficiency before surgery | From the beginning of drug infusion until the moment of starting surgery (assessed up to 30 minutes)
  Respiratory rate < 9/min, Apnea > 29 s, ETCO2 > 54 mmHg, SpO2 < 96%
Respiratory insufficiency during surgery | From the beginning of the surgery until the end of the drug infusion (assessed up to 60 minutes)
  Respiratory rate < 9/min, Apnea > 29 s, ETCO2 > 54 mmHg, SpO2 < 96%

SECONDARY OUTCOMES:
Pain on injection | Just after the beginning of drug infusion
  Patients will answer just after drug infusion begins (Yes or No)
Hypertension | Through the Monitored Anesthetic Care (From the beginning of drug infusion until the end of the drug infusion) up to 60 minutes
  > 140 mmHg during Monitored Anesthetic Care (MAC)
Hypotension | Through the Monitored Anesthetic Care (From the beginning of drug infusion until the end of the drug infusion) up to 60 minutes
  < 90 mmHg during the Monitored Anesthetic Care
Bradycardia | Through the Monitored Anesthetic Care (From the beginning of drug infusion until the end of the drug infusion) up to 60 minutes
  Heart rate < 50/min during the Monitored Anesthetic Care
Tachycardia | Through the Monitored Anesthetic Care (From the beginning of drug infusion until the end of the drug infusion) up to 60 minutes
  Heart rate > 100/min during the Monitored Anesthetic Care
Maximum ETCO2 | Through the Monitored Anesthetic Care (From the beginning of drug infusion until the end of the drug infusion) up to 60 minutes
  ETCO2 will be measured every single respiration in the nasal cavity
Patient satisfaction with Monitored Anesthetic Care | Just before leaving the recovery room
  4-point rating scale on the Satisfaction with MAC
  (4: Fully satisfied, 3: Partially satisfied, 2: Partially unsatisfied,
  1: Totally unsatisfied)
Postoperative Nausea/Vomiting (PONV) | During staying at the recovery room (up to 60 minutes)
  Patients are asked to answer yes/no on PONV, just before leaving the recovery room.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of anesthesiology and pain medicine, Dongguk University Ilsan Hospital, Goyang, Gyeonggido, South Korea

REFERENCES:
- [Background] Zhang X, Li S, Liu J. Correction to: Efficacy and safety of remimazolam besylate versus propofol during hysteroscopy: single-centre randomized controlled trial. BMC Anesthesiol. 2021 Jun 18;21(1):173. doi: 10.1186/s12871-021-01390-x. No abstract available. PMID 34144683
- [Background] Antonik LJ, Goldwater DR, Kilpatrick GJ, Tilbrook GS, Borkett KM. A placebo- and midazolam-controlled phase I single ascending-dose study evaluating the safety, pharmacokinetics, and pharmacodynamics of remimazolam (CNS 7056): Part I. Safety, efficacy, and basic pharmacokinetics. Anesth Analg. 2012 Aug;115(2):274-83. doi: 10.1213/ANE.0b013e31823f0c28. Epub 2011 Dec 20. PMID 22190555
- [Background] Wiltshire HR, Kilpatrick GJ, Tilbrook GS, Borkett KM. A placebo- and midazolam-controlled phase I single ascending-dose study evaluating the safety, pharmacokinetics, and pharmacodynamics of remimazolam (CNS 7056): Part II. Population pharmacokinetic and pharmacodynamic modeling and simulation. Anesth Analg. 2012 Aug;115(2):284-96. doi: 10.1213/ANE.0b013e318241f68a. Epub 2012 Jan 16. PMID 22253270
- [Background] Sneyd JR, Rigby-Jones AE. Remimazolam for anaesthesia or sedation. Curr Opin Anaesthesiol. 2020 Aug;33(4):506-511. doi: 10.1097/ACO.0000000000000877. PMID 32530890
- [Background] Doi M, Morita K, Takeda J, Sakamoto A, Yamakage M, Suzuki T. Efficacy and safety of remimazolam versus propofol for general anesthesia: a multicenter, single-blind, randomized, parallel-group, phase IIb/III trial. J Anesth. 2020 Aug;34(4):543-553. doi: 10.1007/s00540-020-02788-6. Epub 2020 May 16. PMID 32417976